CLINICAL TRIAL: NCT03349229
Title: Description and Evaluation of Care Practices Amongst Geriatric Oncology Unit in the Alpine Valley, in the Follow-up of Cancer Patients.
Brief Title: Geriatric Oncology Follow-up in the Alpine Valley
Acronym: SONGAlp
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC16.058; 2017-A00434-49 (Other: ID RCB)
Record Dates: First submitted 2017-10-13; First posted 2017-11-21 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Oncology; Aging
Keywords: care practices; geriatry; oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As the french population is ageing, the question of medical care in elderly cancer patients is fundamental. A third of all cancer patients are 70 years or older. This population has specific challenges: autonomy maintenance, treatments efficacy with limited side effects.

As a result of a call to projects, the Geriatric Oncology unit of the French Alps (UCOGAlp) has been selected by the National Institute of Cancer (INCa). It includes 15 centres in the Alpine area. This unit has been evaluated patients since 2011, giving them a full geriatric evaluation and trying to establish adapted cares.

In order to evaluate the impact of those evaluation on patients' health, the investigators have developped a geriatric follow-up after 1 month (D30) and 4 months (D120).

The investigators want to develop a common data base to these centres, in order to evaluate the care practices that were developped, and demonstrate the benefit for the patient on the dependence level and the overall survival.

DETAILED DESCRIPTION:
There is a fundamental question nowadays about elderly cancer patients and how investigators can take care of them best. As the French National Institute for cancer stated, a third of all cancers are diagnosed for people over 70 years old. There are specificities for those patients: autonomy maintenance, treatments efficacy with minimum side effects.

This is why the Alpine Unit for Geriatric Oncology (UCOGAlp) was opened, and answered to a national call to projects. It includes 15 hospitals upon the East side of the Rhone-Alpes state. Since 2012, this unit evaluates, according to geriatric oncology validated tests, cancer patients that are 70 years old and older, so they can benefit from an adequate care plan. The need for a geriatric evaluation is determined by the Oncodage test (G8), or on clinical data.

The investigators wanted to see the impact of those initial evaluations, and so the centres developed follow-ups at day 30 and day 120. Investigators want to create a database that gathers the informations from the centres, to evaluate the care practices that were developed, and prove the benefit of such care for the patients, also on physical dependence and overall survival. This will allow new research paths in the field of geriatric oncology.

This study is an observational descriptive one, multicenter, using prospective data for the geriatric oncology as defined by the UCOGAlp.

It is asking the question of registering care practices in several centres of the Alpine valley that have a geriatric consultation, for elderly cancer patients.

The main outcome is the number of follow-ups of patients at 4 months (D120). The secondary outcomes are the adequation between the treatment that is suggested by a committee, the geriatrician's opinion, and the given treatment, the risk factors associated with dependence, and the overall survival.

The patients that are 70 years and older, recently diagnosed with cancer, are included in the study. They have an initial evaluation of their diseases, the autonomy level, a few biological data (hemoglobin, albumen, renal function), other diseases of the patient (and if they have any effect on his autonomy), the treatment that is chosen by specialists. Then there are the follow-ups with the same questions at D30 and D120. The investigators also want to collect data on overall survival after a 2-year follow-up.

The investigators want the analyze from this data to be the start of many projects in geriatric oncology, whether it is for survival or decision of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 70 years old
* Patients diagnosed with cancer (any histologic types)
* Patients amongst the UCOGAlp followup, which includes all patients in the 8 centers that participate

Exclusion Criteria:

* Patients under 70 years old
* Patients with no cancer
* Patients that are not amongst the UCOGAlp followup

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The patients that are recruited for this study are people over 70 years old, recently diagnosed with cancer. They are the patients in the hospitals that usually treat cancer patients. They have to be evaluated by a geriatrician, either after a clinical evaluation, or after they passed an Oncodage G8 test. This test has been validated in France in 2014, then in the international community (Soubeyran et al.). Ths protocole is for all cancer patients, and any cancer localisation. Even if the treatment is only palliative care, the patients can be in the study. The patients have to live in the following countys: Isère, Haute Savoie, Savoie. The participants need to have a geriatric follow up in one of the centers that participates to the SONGAlp study, between January 2013 and December 2017.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of care practices in geriatric oncology | 4 months
  Change in number of geriatric follow ups at D30 and D120

SECONDARY OUTCOMES:
Dependence of the patients | 4 months
  According to a scale of autonomy that is validated , the Instrumental Activities of Daily Living (ranges from 0 to 8/8, o being no abilities to use any instruments and 8 being able to use all kind), and the Activities of Daily Living (0 to 6/6, 0 is being completely depending on others for every day activities like eating or bathing, 6 is being completely autonomous).
Overall survival according to care decisions | 2 years
  We evaluate the mortality for all causes amongst the patients, with subgroups according to the treatment choices

CONTACTS AND LOCATIONS:
Overall Officials: Gaëtan GAVAZZI, PHD, Principal Investigator — CHU Grenoble Alpes; Pascale GUILLEM, PHD, Study Director — CHU Grenoble Alpes
Locations (1):
- CHU Grenoble Alpes, La Tronche, France